CLINICAL TRIAL: NCT01204593
Title: Phase IV, Multicenter, International, Non-comparative, Open Label Study of Efficacy and Safety of Basal Bolus Therapy (Insulin Glargine + Insulin Glulisine) in Patients With T1 Diabetes Previously Uncontrolled on Any Insulin Regimen.
Brief Title: baSal BoluS Therapy in patIenTs With TypE 1 Diabetes Mellitus
Acronym: SUBSTITUTE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_R_05033; U1111-1116-3450 (Other: WHO)
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin glargine + insulin glulisine (Experimental): Insulin glargine dosage will be individually titrated once a week to obtain FPG 80-120 mg/dL (4.5-6.7 mmol/L).
  Insulin glulisine dosage will be individually titrated once a week to obtain a 2-hour postprandial plasma glucose (PPG) < 180 mg/dL (<10.0 mmol/L) and ideally around 140 mg/dL.
  Interventions: Drug: INSULIN GLARGINE; Drug: INSULIN GLULISINE

INTERVENTIONS:
Drug: INSULIN GLARGINE — Pharmaceutical form: solution for injection Route of administration: sub-cutaneous Dose regimen: once a day at bedtime
  Other Names: Lantus SoloStar
Drug: INSULIN GLULISINE — Pharmaceutical form: solution for injection Route of administration: sub-cutaneous Dose regimen: three times a day, preferably just before the meal
  Other Names: Apidra SoloStar

SUMMARY:
Primary Objective:

To evaluate the efficacy of the association Lantus (once-a-day, od) Apidra (thrice-a-day, tid) in terms of change HbA1c from baseline to end of study (week 24), in patients with Type 1 Diabetes Mellitus (T1DM).

Secondary Objectives:

To evaluate:

* The change of hemoglobin A1c (HbA1c) from baseline to week 12
* The percentage of patients with HbA1c < 7% at week 12 and week 24
* The FBG and the 7-point self monitoring of blood glucose (SMBG) at baseline, week 12 and week 24
* The daily dose for both insulin glulisine insulin glargine at baseline, week 12 and week 24
* The incidence of symptomatic hypoglycemias
* Adverse events

DETAILED DESCRIPTION:
After a two-week run-in period patients will enter a six-month treatment period.

Estimated study duration per patient : 26 weeks (including a 2-week run-in period).

ELIGIBILITY:
Inclusion criteria:

1. Known Type 1 diabetic patients (male or female) treated with any type of insulin regimen, except:

   * continuous subcutaneous insulin infusion (CSII, or pump), and
   * patients already treated with insulin glargine
2. Age: 18-60 years inclusive
3. HbA1c: 8% - 10% assessed over the past 6 month
4. At least 1 year of continuous insulin treatment
5. Willingness to accept, and ability to follow:

   * a basal bolus regimen (glargine x1 and glulisine x3 per day),
   * self-monitoring blood glucose (SMBG)
   * a fixed meal plan, or CHO counting
6. Signed informed consent obtained prior to any study procedure

Criteria for entry in the treatment period:

1. HbA1c 8-10% assessed between week -2 and week 0
2. Serum creatinine ≤135 micromol/L in men and ≤110 micromol/L in women
3. Alanine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) lower or equal to three times the upper limit of normal
4. Pregnancy test negative if women of childbearing potential

Exclusion criteria:

1. History of hypersensitivity to insulin glargine and/or insulin glulisine
2. Pregnant, breast-feeding or women of childbearing potential not using efficient contraception
3. Brittle diabetes
4. Known impaired renal function defined as serum creatinine > 135 micromol/L in men and > 110 micromol/L in women at study entry
5. Known impaired hepatic function defined as Alanine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) greater than three times the upper limit of normal at study entry
6. Diabetes ketoacidosis
7. History of drug or alcohol abuse
8. Psychiatric or mental disease
9. Inclusion in another study in the past 6 months or previous inclusion in this study
10. Patient unable or unwilling to manage properly the basal bolus regimen

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 206 (Actual)
Dates: Start 2010-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin A1c (HbA1c) values (following the reference of the International Federation of Clinical Chemistry and Laboratory Medicine (IFCC)) | between baseline (week 0) and endpoint (week 24)

SECONDARY OUTCOMES:
Change of HbA1c | from baseline to week 12
Percentage of patients with HbA1c < 7% | at week 12 and week 24
Fasting Blood Glucose (FBG) | at baseline, week 12 and week 24
7-point Self Monitoring of Blood Glucose (SMBG) | at baseline, week 12 and week 24 (to be performed the week preceding each visit on two consecutive days)
Daily dose for insulin glulisine | At baseline, week 12 and week 24
Daily dose for insulin glargine | At baseline, week 12 and week 24
Symptomatic hypoglycemias | From baseline (week 0) to endpoint (week 24)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (43):
- Algeria (4):
  - Investigational Site Number 01201, Algeries
  - Investigational Site Number 01202, Algiers
  - Investigational Site Number 01203, Algiers
  - Investigational Site Number 01204, Algiers
- Argentina (5):
  - Investigational Site Number 03201, Caba
  - Investigational Site Number 03202, Caba
  - Investigational Site Number 03203, Caba
  - Investigational Site Number 03204, Caba
  - Investigational Site Number 03205, Morón
- Brazil (6):
  - Investigational Site Number 076-007, Curitiba
  - Investigational Site Number 076-003, Distrito Federal
  - Investigational Site Number 076-010, Fortaleza
  - Investigational Site Number 076-006, Marília
  - Investigational Site Number 076-004, Porto Alegre
  - Investigational Site Number 076-002, São Paulo
- Colombia (5):
  - Investigational Site Number 17003, Barranquilla
  - Investigational Site Number 17004, Bogotá
  - Investigational Site Number 17005, Bogotá
  - Investigational Site Number 17007, Bogotá
  - Investigational Site Number 17006, Medellín
- Investigational Site Number 01, Kuwait City, Kuwait
- Mexico (4):
  - Investigational Site Number 48401, Guadalajara
  - Investigational Site Number 48402, Guadalajara
  - Investigational Site Number 48404, Guadalajara
  - Investigational Site Number 48403, Monterrey
- Investigational Site Number 1, Riyadh, Saudi Arabia
- South Africa (12):
  - Investigational Site Number 12468, Benoni
  - Investigational Site Number 710004, Benoni
  - Investigational Site Number 12466, Bloemfontein
  - Investigational Site Number 710006, Bloemfontein
  - Investigational Site Number 12464, Durban
  - Investigational Site Number 12465, Durban
  - Investigational Site Number 710001, Durban
  - Investigational Site Number 710002, Durban
  - Investigational Site Number 12484, Port Elizabeth
  - Investigational Site Number 710003, Port Elizabeth
  - Investigational Site Number 12467, Pretoria
  - Investigational Site Number 710005, Pretoria
- Tunisia (5):
  - Investigational Site Number 78801, Sfax
  - Investigational Site Number 78805, Sfax
  - Investigational Site Number 78803, Tunis
  - Investigational Site Number 78802, Tunis
  - Investigational Site Number 78804, Tunis